CLINICAL TRIAL: NCT01855230
Title: A Randomized, Double-blind, Placebo-controlled, Two-Way Crossover Study to Evaluate the Safety, Tolerability and Clinical Activity of ASM-024 Administered by Dry Power Inhalation to Patients With GOLD 2 (Moderate) or GOLD 3 (Severe) Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Safety, Tolerability, and Clinical Activity of ASM-024 Administered to Patients With GOLD 2 or GOLD 3 Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asmacure Ltée (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ASM-024/II/STA-04
Record Dates: First submitted 2013-05-10; First posted 2013-05-16 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ASM-024

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASM-024 (Experimental): Dry Powder for Inhalation, b.i.d., 14 days
  Interventions: Drug: ASM-024
- Placebo (Placebo Comparator): Dry Powder for Inhalation, b.i.d., 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASM-024 — ASM-024 b.i.d for 14 days
  Arms: ASM-024
Drug: Placebo — Placebo b.i.d. for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and clinical activity of ASM-024 administered as a dry powder for inhalation formulation to patients with GOLD 2 or GOLD 3 COPD.

DETAILED DESCRIPTION:
This is a Phase II, randomized, double-blind, placebo-controlled, two-way crossover study to evaluate the safety, tolerability, and clinical activity of a new, dry powder for inhalation formulation of ASM-024 administered twice daily for 14 days to patients with GOLD-2 or GOLD-3 COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult aged over 40 yrs with a clinically confirmed diagnosis of COPD at the severity stages of GOLD 2 (moderate) or 3 (severe);
* Stable COPD for 1 month prior to screening
* Stable smoker for at least three months prior to screening, or non-smoker, with a smoking history of ≥ 10 packs years;
* FEV₁ ≥ 30 % and < 70 % of the predicted normal value;
* Normal 12-lead ECG

Exclusion Criteria:

* Clinically significant illness except COPD or surgery within 8 weeks prior to first administration of the study medication;
* Significant medical history that, in the Investigator's opinion, may adversely affect participation;
* History of allergy or significant adverse reaction to drugs similar to ASM-024, to nicotine, or to cholinergic drugs or any drugs with a similar chemical structure;
* History of hypersensitivity (anaphylaxis, angioedema) to any drug;
* Positive pregnancy test for female subjects;
* Use of medications known to prolong QT/QTc interval;
* Clinically significant 12 lead ECG at screening;
* Clinically significant physical examination or laboratory findings or abnormal vital signs;
* History of alcohol or drug abuse;
* Positive hepatitis B or C or HIV test at Screening;
* Investigational drug within 30 days of Screening; long-acting investigational drug within 90 days of screening;
* Previous exposure to ASM-024; and
* Women of child-bearing potential and male participants unwilling or unable to use accepted methods of birth control.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
FEV₁ AUC (0 -6 h) | Day 14

SECONDARY OUTCOMES:
Change from baseline in Residual Volume (RV) | Days 1, 2, 3, & 14
Peak change in FEV₁ | Days 1, 2, 3, & 14
Change from baseline in Inspiratory Capacity (IC) | Days 1, 2, 3, & 14
Change from baseline in Functional Residual Capacity (FRC) | Days 1, 2, 3, &14
Change from baseline in FEV₁ | Day 14
Change from baseline in FEV₁/FVC | Days 1, 2, 3, & 14
FVC AUC (0-6 h) | Days 1, 2, 3, & 14
Use of rescue medication | From Day 1 to Day 14

OTHER OUTCOMES:
Safety and Tolerability | Physical examination: Day 14; vital signs: Days 1, 2, 3, & 14; 12-lead ECG: Days 1, 2, 3, & 14; AEs: from Day 1 to patient's final study visit; clinical laboratory evaluations: Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Yvon Cormier, M.D., Study Chair — Asmacure Ltée
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada